# Development and Pilot Testing of an Intervention to Support Interhospital Transfer Decisions (SITe) Regarding Older Adults with Emergency General Surgery Diagnoses

# Documents:

- Pre-intervention SITe survey consent
  - SITe Training Participant Consent

[Note: Consent was obtained through Qualtrics surveys]

9/15/2023

NCT06118359



# **Pre-intervention SITe survey consent**

Angie Ingraham, MD, MS, is inviting you to participate in the Supporting Interhospital Transfer Decisions (SITe) study to understand providers' experiences communicating during calls about interhospital transfers of older (≥60 year old) emergency general surgery patients. This survey should take you about 3 minutes to complete.

Participation is voluntary. You can skip any questions that you cannot or do not want to answer. You can stop at any time.

All answers are confidential and will only be shared with the research team. Results will only be released in aggregate. De-identified data may be kept for future research. The National Institute on Aging, the study funder, may access records pertaining to this research but will not be privy to identifiable information.

The University of Wisconsin-Madison IRB approved this study. If you have any questions about your rights as a research participant or have complaints about the research study or study team, contact the Anonymous Human Research Protection Hotline, which works with research participants to address concerns about research participation and assist in resolving problems. They can be reached at (608)890-1273, (833)652-2506 (toll free), or <a href="https://hrpp@research.wisc.edu">hrpp@research.wisc.edu</a>.

A description of this study will be available on <a href="https://www.clinicaltrials.gov/">https://www.clinicaltrials.gov/</a>. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

For questions related to the study or its results, contact <a href="mailto:egstransferstudy@surgery.wisc.edu">egstransferstudy@surgery.wisc.edu</a>.

By clicking to the next page, you indicate your consent to participate.



# **SITe Training Participant Consent**

Thank you for your interest in the SITe training! Please read the consent information below and select a response.

**Title of Study:** Development and Pilot Testing of an Intervention to Support Interhospital Transfer Decisions (SITe) Regarding Older Adults with Emergency General Surgery Diagnoses

Lead Researcher: Angela Ingraham, MD, MS; email: <a href="mailto:ingraham@surgery.wisc.edu">ingraham@surgery.wisc.edu</a>

#### What is the purpose of this research?

Dr. Angela Ingraham's previous research has shown that communication regarding patients transferred for emergency general surgery (EGS) diagnoses suffers because conversations between referring and accepting providers are ineffective, incomplete, and inefficient. To address this, a group of key stakeholders adapted an existing intervention for interhospital handoffs to address communication surrounding decisions to transfer older EGS patients utilizing extant transfer processes. The purpose of this research is to pilot-test the resulting intervention to Support Interhospital Transfer decisions (SITe) specifically for older EGS patients.

You have been asked to participate because you have engaged in transfer calls of older (≥60 year old) EGS patients.

# Where will the research take place?

This research will be conducted at the University of Wisconsin-Madison (UW). All research activities will take place through secure UW email accounts and web-based seminars.

# What will my participation involve?

Your participation will involve attending a 45-minute virtual seminar to learn about the SITe intervention.

#### Are there any benefits to me?

You are not expected to benefit directly from participating in this study. However, you may experience a benefit from attending the intervention training to learn about improving communication during interhospital transfers of older EGS patients. Also, utilization of the SITe intervention may make the conversations that you have about transfer decisions more effective and efficient.

# Are there any risks to me?

There are minimal risks associated with this research study. A risk of breach of confidentiality always exists; however, we have taken the necessary steps to minimize this risk.

# How will my confidentiality be protected?

To the best of our ability, your participation in this study will remain confidential.



For individuals participating in SITe intervention trainings, the researchers will keep your information confidential and will not share any personal information with anyone outside the research team.

# Will I be paid for participating in this research?

You will be compensated \$100 for attending the SITe intervention training.

### Whom should I contact if I have questions?

You may ask any questions about the research at any time. If you have questions about the research, please contact the Lead Researcher Dr. Angela Ingraham at egstransferstudy@surgery.wisc.edu.

If you have any questions about your rights as a research subject or have complaints about the research study or study team, contact UW Health Patient Relations at 608-263-8009. The Patient Relations Representatives work with research subjects to address concerns about research participation and assist in resolving problems.

Your participation in this research is voluntary, and you may decide not to participate or to withdraw at any time. If you decide not to participate in this study or if you withdraw from participating, you will not be penalized. The results of this study will be used for scholarly purposes. All data is stored in a password protected electronic format on a secure server.

# Please select one of the options below.

- Yes, I consent
- No, I do not consent

| What is your name? |
|--------------------|

Please select the arrow to submit your response. Thank you!